CLINICAL TRIAL: NCT06979180
Title: A Randomized, Triple-blind, Placebo-controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of Papillex® on Abnormal Cervical Cells Caused by HPV
Brief Title: A Clinical Trial to Investigate the Safety and Efficacy of Papillex® on Abnormal Cervical Cells Caused by HPV.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papillex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24PXCFP01
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-05

CONDITIONS: CIN - Cervical Intraepithelial Neoplasia; CIN 1; CIN 2; HPV; Cervical Cells
Keywords: Cervical intraepithelial neoplasia; HPV; Papillex
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papillex® (Experimental): The investigational product, Papillex®, is a dietary supplement containing vitamins B12, C, and E, mixed carotenoids, folate, zinc, selenium, green tea leaf extract, broccoli sprout powder, astragalus, natural all-trans-lycopene and reishi mushroom extracts
  Interventions: Dietary Supplement: Papillex®
- Placebo (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Papillex® — Participants will be instructed to take two capsules twice daily with food, with the first dose taken with the first meal of the day and the second dose taken with the last meal of the day.
  Arms: Papillex®
Other: Placebo — Participants will be instructed to take two capsules twice daily with food, with the first dose taken with the first meal of the day and the second dose taken with the last meal of the day.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of Papillex® on the regression of abnormal cervical cells caused by HPV in women with a cervical intraepithelial neoplasia (CIN) 1 or 2 diagnosis. The main question it aims to answer is:

Is there a difference in the proportion of participants with a regression in CIN based on histology or cytology from baseline at day 180 between Papillex® and placebo?

Participants will be asked to consume Papillex® or placebo for 180 days, complete questionnaires, a PAP smear, HPV test, and colonoscopy (where applicable).

ELIGIBILITY:
Inclusion Criteria:

1. Females between 25 and 55 years of age
2. Females not of child-bearing potential, defined as those who have undergone a permanent sterilization procedure (e.g. hysterectomy, bilateral oophorectomy or bilateral tubal occlusion) or have been post-menopausal for at least 1 year prior to screening Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), hormone implant (Norplant System) or intrauterine hormone-releasing system
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomized partner, provided that partner is the sole sexual partner and that the vasectomised partner has received medical assessment of the surgical success
   * Abstinence
3. Histologically confirmed CIN1+ (as per standard of care) with concordant hrHPV positivity at that time, and current abnormal cytology and hrHPV positivity at screening; interval between historical diagnosis and screening must be >12 months OR documented abnormal cytology (LSIL or worse) plus hrHPV positive >12 months prior, and current abnormal cytology with hrHPV positivity at screening
4. Willing to provide copies of histology and/or cytology reports for eligibility confirmation
5. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
6. Willingness to avoid magnetic resonance imaging, computed tomography, X-ray, or other procedures with contrast media injection for 48 hr prior to study visits assessing micronutrient status
7. Willingness and ability to complete questionnaires and diaries associated with the study, and to complete all clinic visits and assessments
8. Provided voluntary, written, informed consent to participate in the study
9. Otherwise healthy as determined by medical history and laboratory results as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance preventing consumption of investigational product or placebo ingredients
3. Currently undergoing treatment for CIN, are indicated for treatment during the study period, have received treatment (e.g., conization or loop electrosurgical excision procedure) within the last five years, or have active CIN 3
4. Concurrent uterine pathologies
5. History of hysterectomy or destructive therapy of the cervix
6. Cervical cancer
7. Unstable metabolic disease or chronic diseases as assessed by the QI
8. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3)
10. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
11. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
12. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
13. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
14. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
15. Individuals with an autoimmune disease or are immune compromised
16. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
17. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
18. Alcohol intake average of >2 standard drinks per day as assessed by the QI
19. Alcohol or drug abuse within the last 12 months
20. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the investigational product (Section 7.3)
21. Clinically significant abnormal laboratory results at screening as assessed by the QI
22. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
23. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
24. Individuals who are cognitively impaired and/or who are unable to give informed consent
25. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of participants with cytology improvement | Day 0 to 180
  The difference in the proportion of participants with cytology improvement defined as improvement by ≥1 Bethesda category on Pap smear (e.g., HSIL→LSIL/NILM; LSIL→NILM) from baseline at day 180 between Papillex® and placebo.

SECONDARY OUTCOMES:
The difference in the proportion of participants with cytology improvement | Day 0 to 360
  The difference in the proportion of participants with cytology improvement defined as improvement by ≥1 Bethesda category on Pap smear (e.g., HSIL→LSIL/NILM; LSIL→NILM) from baseline at day 360 between Papillex® and placebo.
The difference in the proportion of participants with genotype-specific HPV clearance, | Day 0 to 360
  The difference in the proportion of participants with genotype-specific HPV clearance, defined as negative for the genotypes present at baseline, at day 360 between Papillex® and placebo
Change in immune markers (T lymphocytes, interferon (IFN)-β) between Papillex® and placebo | Day 0 to 180
  Change in immune markers (T lymphocytes, interferon (IFN)-β) from baseline to day 180 between Papillex® and placebo
The difference in the proportion of responders | Day 0 to 180, or 360
  The difference in the proportion of responders, defined as cytology improvement at day 180 OR genotype-specific HPV clearance at day 360
The difference in the proportion of deep responders | Day 0 to 180 and 360
  The difference in the proportion of deep responders, defined as cytology improvement at day 180 AND genotype specific HPV clearance at day 360, between Papillex® and placebo
Concordance between cytology and histology results (where performed as standard of care)* | Day 0 to 360
  Concordance between cytology and histology results (where performed as standard of care)*.
  *For participants who elect to provide colposcopy reports at screening/baseline and during/following completion of the clinical trial (minimum of n = 20; n = 10/group)
Change in micronutrient status | Day 0 to 180
  Change in micronutrient status from baseline to day 180 between Papillex and placebo as assessed by blood concentrations of vitamin B12, folate (vitamin B9), zinc, and selenium.
Change in Symptoms Checklist score between Papillex® and placebo | Day 0 to 180
  Change in Symptoms Checklist score from baseline to days 180 between Papillex® and placebo
Change in Symptoms Checklist score between Papillex® and placebo | Day 0 to 360
  Change in Symptoms Checklist score from baseline to days 360 between Papillex® and placebo
Change in SF-36 Quality of Life (QoL) score between Papillex® and placebo | Day 0 to 180
  Change in SF-36 Quality of Life (QoL) score from baseline to days 180 between Papillex® and placebo
Change in SF-36 Quality of Life (QoL) score between Papillex® and placebo | Day 0 to 360
  Change in SF-36 Quality of Life (QoL) score from baseline to days 360 between Papillex® and placebo
Incidence of post-emergent adverse events (AE) | Day 0 to 360
  Incidence of post-emergent adverse events (AE)

OTHER OUTCOMES:
Clinically relevant changes in blood pressure after supplementation | Day 0 to 180
  Clinically relevant changes in blood pressure after supplementation at Day 180
Clinically relevant changes in heart rate after supplementation | Day 0 to 180
  Clinically relevant changes in heart rate after supplementation at Day 180
Clinically relevant changes in clinical chemistry after supplementation at Day 180 | From enrollment to Day 180
Clinically relevant changes in complete blood count after supplementation at Day 180 | Day 0 to 180

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada